CLINICAL TRIAL: NCT03340636
Title: Relationship Between the Residual Plasma Concentration of Sorafenib and the Occurrence of Adverse Events in Patients Treated for Hepatocellular Carcinoma
Brief Title: Residual Plasma Concentration of Sorafenib and Adverse Events in CHC
Acronym: PharmacoCHC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-109
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Advanced or Metastatic Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, Sorafenib is the only drug therapy to have demonstrated a benefit in overall survival in patients with advanced or metastatic hepatocellular carcinoma. However, this treatment causes many adverse effects that may limit its prescription.

Under these conditions, predicting and therefore potentially preventing the adverse effects of sorafenib is a major issue in the management of patients with hepatocellular carcinoma treated with this drug.

Currently, there is little data available on the correlation between the pharmacokinetics of sorafenib and the side effects of this drug in patients treated for hepatocellular carcinoma.

Investigators propose an observational cohort study evaluating the correlation between residual plasma concentration of sorafenib and the risk of severe adverse effects (grades 3-5) in treatment in patients treated for hepatocellular carcinoma on cirrhosis.

This study should include 60 patients over an expected duration of 12 months. The aim of this work is to determine whether there is a correlation between the residual plasma concentration of sorafenib and the occurrence of severe adverse effects (grades 3-5) at treatment in patients treated for hepatocellular carcinoma on cirrhosis as well as potential influence of the etiology of cirrhosis on this relationship. The ultimate ambition is to be able to anticipate and thus prevent these adverse effects in order to increase the safety of the drug and potentially its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Major Patients.
* Patients with hepatocellular carcinoma on cirrhosis.
* Patients treated for the first time with sorafenib for hepatocellular carcinoma.
* Informed information about the study.

Exclusion Criteria:

* Patients with contraindications to sorafenib.
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with underlying cirrhosis hepatocellular carcinoma treated with Sorafenib
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
residual plasma concentration of sorafenib | from baseline over 6 month
occurrence of severe adverse effects (grades 3-5) | from baseline over 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No